CLINICAL TRIAL: NCT00940810
Title: A Prospective, Randomized, Controlled, Multi Center, Clinical Study With Plasma Disc Decompression Versus Conservative Care
Brief Title: Plasma Disc Decompression Versus Conservative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ArthroCare Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDDCC-001
Record Dates: First submitted 2009-07-15; First posted 2009-07-16 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Decompression, Surgical
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PDD procedure (Experimental)
  Interventions: Procedure: Plasma Disc Decompression/Nucleoplasty
- Conservative Care (Active Comparator)
  Interventions: Procedure: Conservative Care (physiotherapy)

INTERVENTIONS:
Procedure: Plasma Disc Decompression/Nucleoplasty — Subjects assigned to the PDD Group will be scheduled to receive the plasma disc decompression procedure using the Coblation® method.
  Similarly to in Conservative Care group, subjects will be followed-up at 2, 8 weeks, 6 and 12 months (calculated from the date of the PDD procedure). The follow-up visits will consist of a brief physical examination in the clinic and completion of study questionnaires.
  Arms: PDD procedure
Procedure: Conservative Care (physiotherapy) — Subjects assigned to the Conservative Care Group will be scheduled to receive physical therapy according to standard and customary care locally.
  Subjects will be followed-up at 2, 8 weeks, 6 and 12 months . (Calculated from the time of first going through the individual training programme).The follow-up visits will consist of a brief physical examination in the clinic and completion of study questionnaires.
  Arms: Conservative Care

SUMMARY:
The purpose of this study is to compare the plasma disc decompression (PDD) procedure to conservative care (physiotherapy) for the treatment of patients with radicular pain originating from a disc protrusion. Treatment efficacy and rate of improvement is evaluated at 8 weeks after treatment start and followed-up for 1 year after treatment start.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has one symptomatic contained, focal herniated lumbar disc.
2. Patient's age should be at least 18 years old and no more than 65 years old.
3. A VAS score for radicular pain of 50 or greater on a scale of 0 to 100.
4. Radicular pain concordant with image findings (MRI/CT not older than 12 months).
5. Disc height greater or equal to 50% of expected height in the range of a patient's normal anatomic variations and expected changes due to age.
6. Patient signs informed consent.

Exclusion Criteria:

1. Patient is pregnant, or pregnancy is suspected or planned within the study timeframe.
2. Patient has a cardiac pacemaker, automatic defibrillator, or any peripheral stimulator leads in the lumbar area.
3. Allergy to contrast media or drugs to be used in the intended procedure.
4. Medical co-morbidities that preclude surgical intervention.
5. Patient is receiving anti-psychotic therapy.
6. Patient is a prisoner.
7. Patient is incapable of understanding or responding to the study questionnaires.
8. History of previous spinal surgery at, or directly adjacent to, the level to be treated.
9. Patient is morbidly obese (BMI ≥ 40).
10. Patient is simultaneously participating in another device or drug study related to limb/axial pain.
11. Patient has a spinal fracture, tumor or infection.
12. Radicular pain originating from more than one disc level.
13. Axial (back) pain greater than radicular (leg) pain.
14. Clinical evidence of cauda equina syndrome.
15. Progressive neurologic deficit.
16. Radiological evidence of spondylolisthesis at the level to be treated.
17. Radiological evidence of moderate/severe stenosis at the level to be treated.
18. Evidence of extruded or sequestered disc herniation on magnetic resonance imaging.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-08; Primary Completion 2010-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Pain status change assessed using a visual analogue scale (VAS) for radicular pain intensity. | 8 weeks post treatment start

CONTACTS AND LOCATIONS:
Locations (3):
- Raahe Hospital, Raahe, Finland
- Storängskliniken, Stockholm, Sweden
- Pallium Reseach Group; Pain Management, L Ward Seacroft Hospital, Leeds, United Kingdom